CLINICAL TRIAL: NCT01476553
Title: Elimination of Peritoneal Tumor Cells With "Extensive Intraperitoneal Lavage (EIPL)" During Surgical Treatment of Gastric Adenocarcinoma
Brief Title: Elimination of Peritoneal Tumor Cells With Extensive Peritoneal Lavage During Surgery in Patients With Gastric Cancer
Acronym: EIPL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Prematurely halted after interim data analysis
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Principal Investigator, Ulrich Ronellenfitsch, MD, Principal Investigator, Universitätsmedizin Mannheim
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMM-EIPL
Record Dates: First submitted 2011-11-11; First posted 2011-11-22 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Adenocarcinoma; Stomach Neoplasms
Keywords: gastric cancer; extensive intraperitoneal lavage; EIPL; intraperitoneal tumor cells; peritoneal carcinomatosis
MeSH Terms: conditions — Adenocarcinoma; Stomach Neoplasms; Peritoneal Neoplasms | interventions — Therapeutic Irrigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention arm (Experimental): Extensive Intraperitoneal Lavage (EIPL)
  Interventions: Procedure: Extensive Intraperitoneal Lavage (EIPL)

INTERVENTIONS:
Procedure: Extensive Intraperitoneal Lavage (EIPL) — EIPL is performed after completing resection and lymphadenectomy: the abdominal cavity has to be washed ten times with one liter Ringer's solution. Each liter has to be well dispersed manually in the abdominal cavity, and removed and disposed completely. 100 ml of the last liter of lavage fluid will be harvested and sent for analysis.
  Contrary to the Japanese trial, Ringer's solution will be used instead of normal saline solution because of a presumed higher likelihood of peritoneal adhesions when employing the latter (7). Ringer's solution is the standard used for all intraperitoneal lavage procedures at the study centre. To avoid hypothermia, the lavage fluid will be warmed to body temperature (37° Celsius).
  Other Names: EIPL; extensive intraperitoneal lavage; lavage

SUMMARY:
A Japanese study showed that the additional use of an "Extensive Intraperitoneal Lavage" (EIPL), i.e. an extensive washing of the abdominal cavity with water, during surgery for gastric cancer can lead to a significant increase in survival. However, the study was confined to patients in whom upon commencing surgery, free peritoneal tumor cells were detected, which is only a small fraction of patients.

The primary objective of our study is to assess in all patients undergoing removal of the stomach and adjacent lymph nodes for stomach cancer, if EIPL can eliminate free peritoneal tumor cells which have been present at the beginning of the surgery or after the stomach and lymph node removal. Secondary objectives are to assess how often free peritoneal tumor cells occur in patients with stomach cancer, how often surgical resection itself leads to a release of tumor cells, the safety of the EIPL procedure, and disease-free and overall survival of patients undergoing EIPL. Based on the outcome of this japanese study we want to test with special laboratory methods why this lavage leads to a better outcome.

Specifically, the trial will test the hypotheses that a) lymph node dissection causes a release of tumor cells in the abdominal cavity, and b) EIPL eliminates free peritoneal tumor cells.

DETAILED DESCRIPTION:
In spite of the existence of multimodal therapy, the long-term survival of patients with gastric cancer remains poor. In advanced tumor stages, five-year survival rates rarely exceed 30%. One of the factors limiting overall survival is peritoneal carcinomatosis, which frequently occurs after surgical treatment with curative intention.

Peritoneal carcinomatosis is supposed to develop from peritoneal implantation of tumor cells already present in the abdominal cavity during primary surgery. It is assumed that both serosal tumor infiltration and intraoperative lymphadenectomy, which per se leads to a survival improvement (1) and is therefore considered standard in Europe and Japan ((2), http://www.jpca.jp/PDFfiles/ Guidelines2004_eng.pdf), can release tumor cells into the peritoneal cavity. Of note, a Japanese study found that tumor cells were released into the peritoneal cavity during lymphadenectomy in 14-46% of patients, depending on preoperative tumor stage (3).

A randomized clinical trial from Japan (4) demonstrated that an "extensive intraperitoneal lavage" (EIPL), i.e. an irrigation of the abdominal cavity with ten times one liter of physiological saline solution, in combination with intraperitoneal chemotherapy (IPC) carried out after gastrectomy and lymphadenectomy, led to a significant improvement in overall survival compared to patients who received only surgery and IPC without EIPL, and those who received surgery alone without EIPL and IPC. These results suggest that the largest survival benefit is attributable to the addition of EIPL to IPC (5-year survival rate: 43.8% vs. 4.6%) and not to the addition of IPC to surgery alone (5-year survival rate: 4.6% vs. 0%).

However, it is important to consider that the study included only patients in whom peritoneal tumor cells were detected before resection of the stomach and lymph nodes. Thus, only 90 of 1522 (5.9%) patients operated in the participating centers throughout the study period fulfilled the inclusion criteria. Furthermore, the study design was not appropriate to assess if EIPL really leads to a reduction of free tumor cells as assumed. Regarding this hypothesis, the only available results stem from single patients out of smaller studies (4;5). To date, there is no higher level evidence from larger populations.

The present trial, for the first time, uses EIPL as additional treatment in patients with any tumor stage and regardless of the detection of intraperitoneal tumor cells at the beginning of the operation.

Intraperitoneal lavage fluid will be harvested and assessed for tumor cells at three different points of time:

(i) before gastrectomy and lymphadenectomy (ii) after gastrectomy and lymphadenectomy, directly before EIPL (iii) after EIPL

The trial will test the hypotheses that a) lymph node dissection causes a release of tumor cells in the abdominal cavity, and b) EIPL eliminates free peritoneal tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the stomach or cardia (Siewert Type 2 or 3), treated in curative intent with a gastrectomy or subtotal gastrectomy, and D2 lymphadenectomy.
* Adjuvant and neoadjuvant therapy do not constitute exclusion criteria
* Written informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Histologically proven peritoneal carcinomatosis (biopsies of macroscopically suspicious findings must be taken at the beginning of the operation and be analyzed immediately by fresh frozen section)
* Histologically proven distant metastases
* Other medical causes precluding EIPL (e.g. critical condition throughout the surgery with the need to terminate the operation as soon as possible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Peritoneal Conversion Rate (PCR) | intraoperative (day of surgery)
  The Peritoneal Conversion Rate (PCR) is defined as the proportion of patients in whom no free peritoneal tumor cells are detected after EIPL among all patients in whom free peritoneal tumor cells were detected before EIPL. In other words, the PCR measures in what proportion of patients EIPL leads to an elimination of intraperitoneal tumor cells.

SECONDARY OUTCOMES:
Peritoneal Release Rate (PRR) | intraoperative (day of surgery)
  The Peritoneal Release Rate (PRR) is defined as the proportion of patients in whom free peritoneal tumor cells are detected after gastrectomy and lymphadenectomy among all patients in whom no free peritoneal tumor cells were detected before gastrectomy and lymphadnectomy. In other words, this denotes the proportion of patients in whom tumor cells are released into the peritoneal cavity due to the surgical measures performed.
Prevalence of free peritoneal tumor cells before resection | intraoperative (day of surgery)
  This denotes the proportion of patients in whom free intraperitoneal tumor cells can be detected upon laparotomy among all operated patients.
Overall Survival | up to 3 years
  Overall survival is defined as the time between surgery and death, independent of the cause of death.
Recurrence-free survival | up to 3 years
  Recurrence-free survival is defined as the time between surgery and the appearance of a local recurrence, peritoneal carcinomatosis, or distant metastases.
Perioperative in-hospital morbidity | up to the end of the hospital stay (estimated average two weeks after surgery)
  All complications occuring throughout the hospital stay of the patient are assessed according to the Clavien-Dindo classification for surgical complications (6).

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Ronellenfitsch, MD, Principal Investigator — University Hospital Mannheim, Department of Surgery
Locations (1):
- University Hospital Mannheim, Department of Surgery, Mannheim, Germany

REFERENCES:
- [Background] Songun I, Putter H, Kranenbarg EM, Sasako M, van de Velde CJ. Surgical treatment of gastric cancer: 15-year follow-up results of the randomised nationwide Dutch D1D2 trial. Lancet Oncol. 2010 May;11(5):439-49. doi: 10.1016/S1470-2045(10)70070-X. Epub 2010 Apr 19. PMID 20409751
- [Background] Okines A, Verheij M, Allum W, Cunningham D, Cervantes A; ESMO Guidelines Working Group. Gastric cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2010 May;21 Suppl 5:v50-4. doi: 10.1093/annonc/mdq164. No abstract available. PMID 20555102
- [Background] Marutsuka T, Shimada S, Shiomori K, Hayashi N, Yagi Y, Yamane T, Ogawa M. Mechanisms of peritoneal metastasis after operation for non-serosa-invasive gastric carcinoma: an ultrarapid detection system for intraperitoneal free cancer cells and a prophylactic strategy for peritoneal metastasis. Clin Cancer Res. 2003 Feb;9(2):678-85. PMID 12576435
- [Background] Kuramoto M, Shimada S, Ikeshima S, Matsuo A, Yagi Y, Matsuda M, Yonemura Y, Baba H. Extensive intraoperative peritoneal lavage as a standard prophylactic strategy for peritoneal recurrence in patients with gastric carcinoma. Ann Surg. 2009 Aug;250(2):242-6. doi: 10.1097/SLA.0b013e3181b0c80e. PMID 19638909
- [Background] Shimada S, Tanaka E, Marutsuka T, Honmyo U, Tokunaga H, Yagi Y, Aoki N, Ogawa M. Extensive intraoperative peritoneal lavage and chemotherapy for gastric cancer patients with peritoneal free cancer cells. Gastric Cancer. 2002;5(3):168-72. doi: 10.1007/s101200200029. PMID 12378344
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Breborowicz A, Oreopoulos DG. Is normal saline harmful to the peritoneum? Perit Dial Int. 2005 Apr;25 Suppl 4:S67-70. PMID 16300274
- [Derived] Ronellenfitsch U, Ernst K, Mertens C, Trunk MJ, Strobel P, Marx A, Kienle P, Post S, Nowak K. Extensive intraperitoneal lavage to eliminate intraperitoneal tumor cells in gastrectomy with D2 lymphadenectomy for gastric cancer. Tumori. 2018 Oct;104(5):361-368. doi: 10.1177/0300891618792485. Epub 2018 Sep 5. PMID 30185117